CLINICAL TRIAL: NCT06467786
Title: The Therapeutic Effect of Irinotecan Liposomes Combined With Cisplatin/Carboplatin for Platinum Sensitive Recurrent Small Cell Lung Cancer
Brief Title: Study on the Therapeutic Effect of Irinotecan Liposomes in Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202402-30
Record Dates: First submitted 2024-05-28; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Platinum sensitive; Irinotecan liposomes; Second-Line Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental administration group (Experimental): Irinotecan hydrochloride liposome injection: 70mg/m2, intravenous infusion CISPLATIN: 60mg/m2, intravenous infusion or carboplatin: AUC=5, intravenous infusion
  Interventions: Drug: Irinotecan hydrochloride liposome injection

INTERVENTIONS:
Drug: Irinotecan hydrochloride liposome injection — Irinotecan hydrochloride liposome injection combined with platinum

SUMMARY:
This study is a prospective, multicenter, single arm Phase II exploratory study. It is expected to include 24 first-line patients with small cell lung cancer who have progressed after 6 months of treatment with platinum containing regimens, and receive treatment with irinotecan liposomes combined with cisplatin or carboplatin regimens.

DETAILED DESCRIPTION:
Based on literature research and the birth of independently developed irinotecan liposomes by Shiyao, we plan to conduct a therapeutic study on the combination of irinotecan liposomes and cisplatin/carboplatin for platinum sensitive recurrent small cell lung cancer. The aim is to explore the efficacy and safety of the combination of irinotecan liposomes and platinum based chemotherapy regimen in first-line treatment of small cell lung cancer patients who have progressed after 6 months using platinum based regimens, providing better clinical evidence for use.

The research unit is the Second Affiliated Hospital of Air Force Military Medical University. The study includes screening period (within 28 days), treatment period, and follow-up period (safety follow-up and PFS follow-up). The subjects signed an informed consent form and underwent baseline examination during the screening period. Patients who met the inclusion and exclusion criteria entered the treatment period. All subjects completed the relevant examinations specified in the protocol during the treatment process to observe safety, tolerance, and efficacy. The same subject only received one dosing plan during the study period. After the treatment period ends, enter the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The patient fully understands this study, voluntarily participates and signs an informed consent form (ICF).
* Age ≥ 18 years old;
* Patients with extensive stage small cell lung cancer diagnosed by pathology or histology;
* According to RECIST 1.1 standard, patients have at least one measurable target lesion; For lesions that have undergone radiation therapy in the past, they can only be included as measurable lesions if there is clear disease progression after radiation therapy;
* Progression confirmed by imaging examination after 6 months of first-line radiotherapy and chemotherapy containing platinum drugs or platinum regimen radiotherapy and chemotherapy ± immunotherapy;
* Eastern Cancer Collaborative Group (ECOG) physical fitness score: 0-2 points;
* Estimated survival time ≥ 3 months;
* Absolute neutrophil count (ANC) ≥ 1.5 x 10 ^ 9/L, platelet count ≥ 90 x 10 ^ 9/L, and hemoglobin count ≥ 90 g/L (no blood transfusion, blood products, use of granulocyte colony-stimulating factor or other hematopoietic stimulating factor correction within 14 days prior to laboratory examination);
* Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of normal value; AST and ALT ≤ 2.5 times the upper limit of normal values (≤ 5 times the upper limit of normal values for patients with liver invasion); Total bilirubin ≤ 1.5 times the upper limit of normal value (≤ 3 times the upper limit of normal value for patients with liver invasion);
* Women of childbearing age must undergo a pregnancy test (serum) within 7 days before enrollment, and the result is negative. They are willing to use appropriate methods of contraception during the trial period and 6 months after the last administration of the trial drug;

Exclusion Criteria:

* Patients with large cell neuroendocrine tumors and mixed small cell carcinoma;
* Patients with active brain metastasis or central nervous system invasion confirmed by imaging evaluation and/or biopsy (prednisone equivalent dose ≥ 10mg);
* There is an hypersensitivity reaction to any investigational drug or its components;
* Severe uncontrolled concurrent infections or other serious uncontrolled concomitant diseases, moderate or severe kidney injury; (such as progressive infection, uncontrollable hypertension, diabetes, etc.);
* Heart function and disease meet one of the following conditions:

  1. Long QTc syndrome or QTc interval>480 ms;
  2. Complete left bundle branch block, II or III degree atrioventricular block;
  3. Severe and uncontrolled arrhythmias that require medication treatment;
  4. The New York College of Cardiology has a classification of ≥ III;
  5. Cardiac ejection fraction (LVEF) below 50%;
  6. A history of myocardial infarction, unstable angina, severe unstable ventricular arrhythmias, or any other arrhythmias requiring treatment, a history of clinically severe pericardial disease, or evidence of acute ischemic or active conduction system abnormalities on electrocardiogram within the 6 months prior to recruitment.
* Active infection of hepatitis B and hepatitis C (hepatitis B B virus surface antigen is positive and hepatitis B B virus DNA exceeds 1x103 copies/mL; hepatitis C virus RNA exceeds 1x103 copies/mL);
* Human Immunodeficiency Virus (HIV) infection (HIV antibody positive);
* Has previously or currently suffered from other malignant tumors (except for effectively controlled non melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have not been treated and have been effectively controlled within the past five years);
* Pregnant and lactating women, as well as patients of childbearing age who are unwilling to take contraceptive measures;
* Patients with other malignant tumors that require treatment; The researchers determined that patients who are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective response rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 1 years.
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with response of Complete Response or Partial Response, will be assessed up to 1 years.

SECONDARY OUTCOMES:
Progression-free survival | Progression-free survival (PFS) analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 4 years
  Progression free survival (PFS) refers to the time from recording the first chemotherapy treatment to the date of disease progression, as assessed by researchers.
Duration of Response | Duration of Response（DoR）analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 4 years
  Duration of Response（DoR）refers to the time from the first assessment as CR or PR to the first assessment as PD or (due to any reason) death
Overall Survival | The maximum time from receiving treatment to dying for any reason is 4 years.
  Overall survival (OS) refers to the time that researchers evaluate from recording the first chemotherapy to death (of any cause).
Safety/Adverse event | From the first recorded chemotherapy to 4 weeks after the last recorded chemotherapy
  Incidence of Adverse Events (AEs): Incidence, severity and seriousness of adverse events, incidence of serious adverse events (SAEs), which usually be graded by CTCAE v5.0 based on current clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Haichuan Su, PhD, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No